CLINICAL TRIAL: NCT00181116
Title: Efficacy of Levetiracetam for Language Dysfunction Associated With Benign Epilepsy With Centrotemporal Spikes
Brief Title: Levetiracetam for Benign Rolandic Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-02-18-06
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Epilepsy
Keywords: Epilepsy; Benign rolandic; Levetiracetam
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam

SUMMARY:
This study is designed to test if the language problems commonly seen in children with benign rolandic epilepsy would improve by switching anticonvulsants to levetiracetam.

DETAILED DESCRIPTION:
This is a 6 month study in which children on another anticonvulsant would have EEG, language testing, and a clinic visit at baseline. They would then be rapidly transitioned off of their current anticonvulsant and onto levetiracetam (Keppra). Repeat EEG and language testing would be done after 6 months to evaluate for improvement.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6-12
* Benign rolandic epilepsy
* Language difficulties as reported by parents or teachers
* On another anticonvulsant other than levetiracetam

Exclusion Criteria:

* Prior use of levetiracetam
* On 2 or more anticonvulsants
* Language problems prior to epilepsy
* Another seizure disorder
* Status epilepticus within the past 6 months
* Significant psychiatric disease
* Progressive neurologic disease

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6
Dates: Start 2005-03; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Language improvement

SECONDARY OUTCOMES:
Seizure control

CONTACTS AND LOCATIONS:
Overall Officials: Eric H Kossoff, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Bello-Espinosa LE, Roberts SL. Levetiracetam for benign epilepsy of childhood with centrotemporal spikes-three cases. Seizure. 2003 Apr;12(3):157-9. doi: 10.1016/s1059-1311(03)00004-9. PMID 12651081
- [Background] Kossoff EH, Boatman D, Freeman JM. Landau-Kleffner syndrome responsive to levetiracetam. Epilepsy Behav. 2003 Oct;4(5):571-5. doi: 10.1016/s1525-5050(03)00171-9. PMID 14527502